CLINICAL TRIAL: NCT07185035
Title: An Exploratory Clinical Study on the Safety and Efficacy of Autologous NK Cells in the Treatment of Pulmonary Nodules
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Rui Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-089
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Nodules, Solitary; Pulmonary Nodules, Multiple
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN5001 (Experimental)
  Interventions: Biological: KN5001

INTERVENTIONS:
Biological: KN5001 — Subjects will receive KN5001 on day0, 3, and 6. Multiple Doses of KN5001 will infused using the "3 + 3" dose-escalation strategy.

SUMMARY:
A single-center, open-label dose-escalation design to evaluate the safety and efficacy of KN5001 in patients with pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily sign the informed consent form, understand this clinical study, and are willing to follow and able to complete all trial procedures;
2. 18-70 years old, male or female;
3. Subjects with lung nodules confirmed by imaging examination must meet the following conditions:

   Multiple high-risk nodules have been surgically removed and confirmed to be malignant lesions, and the remaining high-risk nodules (refer to the standards in Appendix 12) cannot be surgically removed again, and are not suitable for other effective treatments or have failed other treatments;
4. If the subject is unable to complete the puncture or the puncture fails, the subject must be diagnosed as a malignant nodule through PET-CT imaging examination.

Exclusion Criteria:

1. Subjects who are known to have allergic reactions, hypersensitivity reactions, intolerances or contraindications to any component of KN5001, or subjects with a history of severe allergic reactions;
2. Subjects with the following genetic syndromes: Fanconi syndrome, Kostmann syndrome, Shwachman syndrome or any known bone marrow failure syndrome;
3. Subjects with active or uncontrolled infections requiring parenteral antibiotics; Evidence of a serious active viral or bacterial infection or an uncontrolled systemic fungal infection;
4. Subjects with heart failure of grade III or IV according to the New York Heart Association (NYHA) cardiac function classification standard (see Appendix 1);
5. Subjects with a history of epilepsy or other central nervous system diseases;
6. Subjects with a history of malignant tumors, excluding patients with cured skin or cervical carcinoma in situ and patients with inactive tumors;
7. Subjects with a significant bleeding tendency, such as gastrointestinal bleeding, coagulopathy, hypersplenism, etc.;
8. Subjects with unstable angina, symptomatic congestive heart failure, or myocardial infarction in the past 6 months;
9. Females who are pregnant, lactating, or planning a pregnancy within six months;
10. Subjects who have received other clinical trial treatment within 3 months;
11. Any situation judged by the investigators that may increase the risk of the subjects or interfere with the clinical trial outcome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of all adverse events occurring within 28 days after the first infusion of KN5001 | Time Frame: up to 28 days after infusion
  To characterize the Treatment Emergent Adverse Events (TEAEs) of KN5001 for patients with pulmonary nodules

SECONDARY OUTCOMES:
The overall response rate (ORR) | Time Frame: 6 and 12 months after infusion
  To characterize the efficacy of KN5001 for patients with pulmonary nodules
Disease control rate (DCR) | Time Frame: 6 and 12 months after infusion
  To characterize the efficacy of KN5001 for patients with pulmonary nodules

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No